CLINICAL TRIAL: NCT03277872
Title: NoL Index, Heart Rate and Mean Arterial Blood Pressure Responses to Tracheal Intubation Performed With MacIntosh Blade Versus Glidescope
Brief Title: NoL, HR and MABP Responses to Tracheal Intubation Performed With MAC Blade Versus Glidescope
Acronym: NoLint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Verathon (Industry); Canadian Hospital Specialties Ltd (Unknown)
Responsible Party: Principal Investigator, Philippe Richebe, Principal Investigator, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-1144
Record Dates: First submitted 2017-08-29; First posted 2017-09-11 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Intubation; Nociceptive Pain; Anesthesia; Laryngoscopy
MeSH Terms: conditions — Nociceptive Pain | interventions — Laryngoscopy

STUDY DESIGN:
Intervention Model Description: In this study, each patient will be exposed to three laryngoscopies; one with the single use blade for the GlideScope and without ETT; one with the Macintosh laryngoscopy and without ETT; and one with the ETT insertion (laryngoscopy done with either GlideScope or Macintosh according to second randomization). The order in which will be used either the GlideScope or the MAC blade for the first two laryngoscopies will be decided according to the first randomization.
  This will lead to 2 different groups for the first randomization process regarding our primary objective:
  * GVL / MAC-DL / GVL or MAC-DL+ETT,
  * MAC-DL / GVL / GVL or MAC-DL+ETT.
  The tool used for the third laryngoscopy will be decided according to a second randomization, necessary to one of our secondary objectives.
  Each patient will be its own control when comparing nociceptive response to different laryngoscopy/intubation tool (no need for control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GlideScope (GVL) Blade (Active Comparator): Patients in this arm will have the first laryngoscopy performed with the GlideScope (GVL) blade and the second one with the MacIntosh blade. The tool used for the third laryngoscopy, followed by intubation, (either GlideScope or MAC blade) will be decided according to a second randomization, necessary to one of our secondary objectives.
  Interventions: Device: Laryngoscopy with GlideScope (GVL) Blade
- MacIntosh (MAC) Blade (Active Comparator): Patients in this arm will have the first laryngoscopy performed with the MacIntosh (MAC) blade and the second one with the GlideScope blade. The tool used for the third laryngoscopy, followed by intubation, (either GlideScope or MAC blade) will be decided according to a second randomization, necessary to one of our secondary objectives.
  Interventions: Device: Laryngoscopy with MacIntosh (MAC) Blade

INTERVENTIONS:
Device: Laryngoscopy with GlideScope (GVL) Blade — 1. st Laryngoscopy with GVL Blade
  2. nd Laryngoscopy with MAC Blade
  3. rd Laryngoscopy and ETT insertion with either GVL or MAC Blade according to 2nd randomization
  Arms: GlideScope (GVL) Blade
Device: Laryngoscopy with MacIntosh (MAC) Blade — 1. st Laryngoscopy with MAC Blade
  2. nd Laryngoscopy with GVL Blade
  3. rd Laryngoscopy and ETT insertion with either GVL or MAC Blade according to 2nd randomization
  Arms: MacIntosh (MAC) Blade

SUMMARY:
Prospective, randomized and controlled who will be conducted in Maisonneuve-Rosemont hospital and whose objectives are:

* To observe if the alterations of the NoL index and the standard monitoring (Mean Arterial Blood Pressure and Heart Rate) (using the variability of NoL index and standard monitoring, peak NoL index and peak standard monitoring values, and number of time passed over their respective threshold for nociceptive response) are more accentuated after laryngoscopy using the classical MAC blade versus single-use disposable blade of the Glidescope.
* To observe the nociceptive response (using the variability of NoL index and standard monitoring, peak NoL index and peak standard monitoring values, and number of time passed over their respective threshold for nociceptive response) related to the insertion of endotracheal tube between vocal cords during the intubation.

Study plans to enroll 50 adult patients scheduled to undergo either general, gynecological, neurological, orthopedic, plastic or urological surgery under general anesthesia and who necessitate endotracheal intubation.

DETAILED DESCRIPTION:
The purpose of this prospective pragmatic study is to evaluate the changes in NoL index, Heart Rate (HR) and Mean Arterial Blood Pressure (MABP) following the painful stimulus that represents laryngoscopy and intubation performed using either the single use blade of the Glidescope (group GVL) or the classically used MAC blade (group MAC). Calculation will be using the variations of NoL, HR and MABP, the peak values of these 3 parameters, and also the area above the curve of each parameter for 3 minutes (above the mean pre-stimulus values) and the amount of time (out of 3 minutes post-stimulus) those 3 parameters will be significantly higher than their respective pre-intubation mean thresholds.

In this prospective, randomized and controlled study, each patient will normally enter the operating room on the day of his surgery. All the normal monitors are installed, along with the NoL monitor. Pre-oxygenation (with 100% 02) is then started. While the patient is doing the pre-oxygenation, MABP, HR and NoL index measures are gathered to establish a baseline for each patient.

Once pre-oxygenation is over, induction with xylocaïne, propofol, remifentanil and rocuronium is given (according to patients' ideal weight). The end of the remifentanil bolus will correspond to the time 0 of our study. To be sure our patients are sleeping and on the same level of anesthetic medication during our study, perfusions of propofol and remifentanil will be administred until tracheal intubation and inhaled anesthetic gaz given. When the patient is asleep and apneic, a Guedel device (chosen according to patient weight and height) is inserted in the mouth, as in usual practice, to ease the manual ventilation until the laryngoscopy. The patient is then ventilated with a face mask. After 5 minutes, the first laryngoscopy is performed (either with GlideScope blade or MAC blade according to randomization). Once a Cormack-Lehane grade I or II is obtained, the movement is ended, and the patient is ventilated again for 4 minutes with the Guedel. If the procedure takes more than 30 seconds to perform (if no view of grade I or II is seen before 30 seconds), the laryngoscopy is considered difficult and the patient will be excluded from the study. At T9 (9 minutes after T0), the second laryngoscopy is done (either with the MacIntosh blade or the GVL blade - the tool used for the second laryngoscopy will always be the one that wasn't used at the first laryngoscopy). The size of the MacIntosh blade (MAC 3 or 4) or the disposable blade for GVL is decided according to the patient size (height and weight). At the second laryngoscopy, the endotracheal tube is still not inserted, only the procedure of laryngoscopy is done, so that we can evaluate the hemodynamic and the NoL index responses related only to the type of device used for laryngoscopy. Then, the operator replaces the Guedel and ventilates the patient with a facemask (100% O2) for 4 more minutes, without stimulating the patient otherwise. At T13 (13 minutes after T0), the third laryngoscopy will be performed (either with the single-use blade for GlideScope or the MacIntosh blade - according to randomization). This time, the ETT is inserted (size 7 or 8, depending on the size and sex of the patient). After ETT insertion, the patient is then ventilated with the anesthesia machine and the perfusions of propofol/remifentanil is discontinued.

Monitors will record HR, MABP and NoL index until 3 minutes after the ETT insertion (end of the study). All the data will be electronically registered every 5 seconds and exported in an anonymous manner for each patient into an excel file at the end of the study.

In this study, each patient is exposed to three laryngoscopies; one with the single use blade for the GlideScope, one with the Macintosh laryngoscopy and one with the ETT insertion (laryngoscopy done with either GlideScope or Macintosh according to randomization). Hence, each patient will be its own control. It will then be more reliable to compare the differences in nociceptive response according to the tool used for laryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I or II
* Mallampati class I or II
* Patients > 18 years old
* Elective general, gynecological, neurological, orthopedic, plastic or urological surgery under general anesthesia
* Type of surgery that usually necessitate endotracheal intubation and controlled ventilation

Non-inlusion Criteria:

* Patient refusal
* History of psychiatric diseases or psychological problems (including mental retardation); inability to give consent; language barrier.
* Anticipated difficult airway (Mallampati class III and IV, thyromental distance < 6 cm, mouth opening < 3 cm, neck extension <80° and neck flexion <35°, inability to prognath, meaning bringing lower mandibular before the upper maxilla)
* Patient with history of neck rigidity or instability
* BMI > 30
* Patient with beard (because of recognized risk for difficult ventilation)
* Patient with history of oropharyngeal or tracheal surgery (excluding adenoidectomy, amygdalectomy and teeth removal)
* Severe coronary artery disease
* Serious cardiac arrhythmias (including atrial fibrillation)
* Use of β-blockers (all types)
* History of opioid or illicit drug substance abuse
* Chronic use of psychotropic and/or opioid drugs
* Allergy to remifentanil or propofol
* Pregnancy
* Contraindications to mask ventilation (GI tract obstruction, pregnancy, active GERD, non-fasting patients)
* Difficult mask ventilation (before randomization at the first laryngoscopy)

Exclusion Criteria:

* Unexpected difficult airway requesting excessive, possibly painful airway manipulations
* Requiring hemodynamic support with vasopressors or inotropes 5 minutes before first laryngoscopy to 3 minutes after insertion of ETT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Delta NoL | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the variation of NoL (delta NoL) after laryngoscopy using the single use blade for Glidescope (GVL) versus MAC blade (MAC) in anesthetized patients

SECONDARY OUTCOMES:
Delta Heart Rate | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the variation of the standard hemodynamic parameter after laryngoscopy using the single use blade for Glidescope (GVL) versus MAC blade (MAC) in anesthetized patients
Delta Mean Arterial Blood Pressure | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the variation of the standard hemodynamic parameter after laryngoscopy using the single use blade for Glidescope (GVL) versus MAC blade (MAC) in anesthetized patients
Peak value of NoL | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the peak value of NoL after laryngoscopy in the GVL group versus the MAC group
Peak value of Heart Rate | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the peak value of standard hemodynamic parameter after laryngoscopy in the GVL group versus the MAC group
Peak value of Mean Arterial Blood Pressure | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the peak value of standard hemodynamic parameter after laryngoscopy in the GVL group versus the MAC group
Amount of time (in seconds) Mean Arterial Blood Pressure is over its baseline value after laryngoscopy stimulus | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the amount of time (in seconds) the MABP will spend over its respective mean pre-stimulus value after laryngoscopy with GVL versus MAC
Amount of time (in seconds) NoL, is over its baseline value after laryngoscopy stimulus | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the amount of time (in seconds) the NoL will spend over its respective mean pre-stimulus values after laryngoscopy with GVL versus MAC
Amount of time (in seconds) Heart Rate is over its baseline value after laryngoscopy stimulus | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the amount of time (in seconds) the HR will spend over its respective mean pre-stimulus value after laryngoscopy with GVL versus MAC
Area Under the Curve for NoL for GVL versus MAC blade | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the area under the curve between GVL versus MAC-Dl laryngoscopy that NoL spends above its baseline value and calculated for the 3 minutes after the stimulus
Area Under the Curve for Heart Rate for GVL versus MAC blade | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the area under the curve between GVL versus MAC-Dl laryngoscopy that HR spends above its baseline value and calculated for the 3 minutes after the stimulus
Area Under the Curve for Mean Arterial Blood Pressure for GVL versus MAC blade | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the area under the curve between GVL versus MAC-Dl laryngoscopy that MABP spends above its baseline value and calculated for the 3 minutes after the stimulus
Variation of NoL for laryngoscopy versus laryngoscopy + endotracheal intubation | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the variation of NoL after the laryngoscopy alone versus laryngoscopy + endotracheal tube (ETT) insertion in the GVL and the Mac group
Variation of HR for laryngoscopy versus laryngoscopy + endotracheal intubation | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the variation of HR after the laryngoscopy versus laryngoscopy + endotracheal tube (ETT) insertion in the GVL and the Mac group
Variation of MABP for laryngoscopy versus laryngoscopy + endotracheal intubation | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the variation of MABP after the laryngoscopy versus laryngoscopy + endotracheal tube (ETT) insertion in the GVL and the Mac group
Peak value of NoL for laryngoscopy versus laryngoscopy + endotracheal intubation | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the peak value of NoL after the laryngoscopy + endotracheal tube (ETT) insertion in the GVL and the Mac group
Peak value of HR for laryngoscopy versus laryngoscopy + endotracheal intubation | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the peak value of HR after the laryngoscopy + endotracheal tube (ETT) insertion in the GVL and the Mac group
Peak value of MABP for laryngoscopy versus laryngoscopy + endotracheal intubation | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the peak value of MABP after the laryngoscopy + endotracheal tube (ETT) insertion in the GVL and the Mac group
Area Under the Curve of NoL for laryngoscopy versus laryngoscopy + endotracheal intubation | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the AUC of NoL after the laryngoscopy + endotracheal tube (ETT) insertion in the GVL and the Mac group
Area Under the Curve of HR for laryngoscopy versus laryngoscopy + endotracheal intubation | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the AUC of HR after the laryngoscopy + endotracheal tube (ETT) insertion in the GVL and the Mac group
Area Under the Curve of MABP for laryngoscopy versus laryngoscopy + endotracheal intubation (with both devices) | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the AUC of MABP after the laryngoscopy + endotracheal tube (ETT) insertion in the GVL and the Mac group
Delta NoL analyzed according to order of randomization to see if this order influences its response | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the influence of the order of the tool used for laryngoscopies with the variation of NoL, after laryngoscopy using the single use blade for Glidescope (GVL) and MAC blade (MAC) in anesthetized patients
Delta Heart Rate analyzed according to order of randomization to see if this order influences its response | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the influence of the order of the tool used for laryngoscopies with the variation of HR, after laryngoscopy using the single use blade for Glidescope (GVL) and MAC blade (MAC) in anesthetized patients
Delta Mean Arterial Blood Pressure analyzed according to order of randomization to see if this order influences its response | From 30 seconds before to 3 minutes after each laryngoscopy (3 total) for each patient
  To compare the influence of the order of the tool used for laryngoscopies with the variation of MABP, after laryngoscopy using the single use blade for Glidescope (GVL) and MAC blade (MAC) in anesthetized patients

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Richebe, MD, PhD, Principal Investigator — Université de Montréal
Locations (1):
- Hopital Maisonneuve Rosemont, CIUSSS de l'Est de l'Ile de Montreal, Montreal East, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sbeghen V, Verdonck O, McDevitt J, Zaphiratos V, Brulotte V, Loubert C, Tanoubi I, Drolet P, Belanger ME, Fortier LP, Godin N, Guertin MC, Fortier A, Richebe P. A randomized controlled trial comparing nociception level (NOL) index, blood pressure, and heart rate responses to direct laryngoscopy versus videolaryngoscopy for intubation: the NOLint project. Can J Anaesth. 2021 Jun;68(6):855-867. doi: 10.1007/s12630-021-01936-0. Epub 2021 Mar 11. PMID 33709262